CLINICAL TRIAL: NCT05656092
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Phase III Study to Evaluate the Efficacy and Safety of HIP0612 in Patients With Gastric Ulcer
Brief Title: A Study to Evaluate the Effiacy and Safety of HIP0612 in Patients With Gastric Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-AESOP-301
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Gastric Ulcer
MeSH Terms: conditions — Stomach Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIP0612 (Experimental): Taking HIP0612+HPP2202 once daily for 4 or 8 weeks.
  Interventions: Drug: HIP0612; Drug: HPP2202
- RLD2204 (Active Comparator): Taking RLD2204+HPP2201 once daily for 4 or 8 weeks.
  Interventions: Drug: RLD2204; Drug: HPP2201

INTERVENTIONS:
Drug: HIP0612 — Test drug
  Arms: HIP0612
Drug: HPP2202 — Placebo drug
  Arms: HIP0612
Drug: RLD2204 — Reference drug
  Arms: RLD2204
Drug: HPP2201 — Placebo drug
  Arms: RLD2204

SUMMARY:
A multicenter, randomized, double-blind, active-controlled, phase III study to evaluate the efficacy and safety of HIP0612 in patients with gastric ulcer.

ELIGIBILITY:
Inclusion Criteria:

* 19 years to 75 years
* Diagnosis of active gastric ulcers according to the Sakita-Miwa classification from upper GI endoscopy
* Patients understood the consents and purpose of this trial and signed consent form

Exclusion Criteria:

* Patients who cannot perform endoscopy
* Finding of malignancy, duodenal ulcer, ulcer perforation, postoperative (eg, endoscopic mucosal resection, endoscopic submucosal dissection) ulcer(s), Barrett's oesophagus measuring >3cm, oesophageal dysplasia, oesophageal and/or gastric varices, bleeding disorder on upper GI endoscopy
* History of definitive acid lowering surgery or pervious oesophageal or gastric surgery (except for benign tumor excisionn, simple close of perforations)
* Zollinger-Ellison syndrome, pyloric stenosis, oesophageal motility disorder, esophageal stricture
* Severe hepatic disease
* Severe renal disease, CKD
* Bleeding disorder
* History of malignancy or was treated for malignancy within 5 years before the start of the Visit 1
* Patients who have taken drugs containing following list within 2 weeks prior to upper GI endoscopy, or requirement of persistent use of drugs during the study period: acid suppressive drugs, antacids, anticholinergic drugs, gastroprotective agent
* Patients who have taken drugs containing following list within 1 weeks prior to upper GI endoscopy, or requirement of persistent use of drugs during the study period: antithrombotic agents, NSAIDs, aspirin
* Requirement of use of excluded medications during the study
* History of allergic reaction to the medications used in this study
* Glucose-galactose malabsorption, Fructose intolerance, Sucrase-isomaltase deficiency
* Use of other investigational drugs within 30 days prior to the study
* History of alcohol or drug abuse
* Positive to pregnancy test, nursing mother, intention on pregnancy
* Considered by investigator as not appropriate to participate in the clinical study with other reason

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Healing rate of gastric ulcer | week 8
  Including subjects endoscopically confirmed healing of gastric ulcer after 4 Weeks of treatment and complete the study

SECONDARY OUTCOMES:
Healing rate of gastric ulcer | week 4
Healing rate of gastric ulcer according to H.pylori infection status | week 4, 8
Post-treatment resolution rate of GI symptoms | week 4, 8

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No